CLINICAL TRIAL: NCT05924204
Title: Effect of Photobiomodulation on Pain Control After Placement of Elastomeric Spacers: a Randomized Controlled Trial.
Brief Title: Effect of Photobiomodulation on Pain Control After Placement of Elastomeric Spacers.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INFLAURU
Record Dates: First submitted 2023-06-18; First posted 2023-06-29 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1 TREATMENT GROUP (Experimental): In the Treatment group the FMB with 4 J of energy by point
  Interventions: Radiation: Photobiomodulation
- G2 SHAM GROUP (Sham Comparator): In the Sham group, the the device will be turned off
  Interventions: Other: Simulation of Photobiomodulation

INTERVENTIONS:
Radiation: Photobiomodulation — Application of photobiomodulation
  Arms: G1 TREATMENT GROUP
Other: Simulation of Photobiomodulation — Simulation of photobiomodulation
  Arms: G2 SHAM GROUP

SUMMARY:
Recent studies have shown that photobiomodulation (FBM) can modulate pain after the placement of elastomeric separators, however, to date, there is no ideal protocol for its application. Therefore, the objective of this study will be to evaluate the effect of photobiomodulation on pain control 24 hours after the placement of elastomeric separators using the visual analog scale (VAS). 25 patients between 13 and 30 years old with the need for the placement of orthodontic bands in the lower first molars bilaterally will be included, which establishes a sample of fifty molars.

Elastomeric separators will be placed on the mesial and distal surfaces of the right and left molars. Treatment will be randomized to the right molar and the opposite treatment will be applied to the left side. The study groups will be G1 (experimental) - elastomeric separators + FBM (diode laser, 808nm, 100mw power, with 2 J, 3 points per vestibular and 3 points per palatal, single session, 707J/cm2) and G2-(control)- elastomeric separators + FBM simulation. The patient and the evaluator will be blinded to the intervention performed. The primary outcome variable will be spontaneous pain assessed 24 hours after the placement of elastomeric separators measured with the VAS scale. Secondary outcome variables will be pain during mastication (measured with the VAS scale), count of the number of analgesics (paracetamol), local temperature (measured with a digital thermometer), and assess the impact of oral health on quality of life. of the participant, the OHIP-14 questionnaire will be applied. These outcomes will be evaluated at baseline, 24 with the presence of the participant, and 72 hours after the placement of elastomeric separators. If the data are normal, they will be submitted to the ANOVA - one-way test. Data will be presented as means ± SD and the p-value will be set to < 0.05.

DETAILED DESCRIPTION:
This randomized, controlled, double-blind, split-mouth clinical trial meets the criteria for designing a clinical study under the conditions of the SPIRIT Statement. The study was approved by the Committee for Ethics in Research (CEP) of the Universidad Católica del Uruguay. The participants who will be recruited are patients who are undergoing orthodontic treatment at the Orthodontic Clinic of the Specialization Course in Orthopedics and Orthodontics at the Catholic University of Uruguay in the city of Montevideo, Uruguay; those who require the installation of bands on the lower first permanent molars.

Any change or change will be reported and clarified to the CEP and informed in publications. A copy of the signed informed consent will be sent to the participant by email (completed in the TCLE). The project will be registered at www.clinicaltrial.gov There is no conflict of interest about any product used in the work and about any author involved in the studio. The data will be published and there will be no restriction on the inclusion of data for publication. All data will be available for your consultation, and all patients will have access to their medical records at any time they wish.

ELIGIBILITY:
Inclusion Criteria:

* Patients will include:

  * With the need to place bilateral orthodontic bands on the lower first molars.
  * Age 13 to 30 years old.
  * Both sexes.
  * No comorbidities.
  * Never used orthodontic appliances.
  * Preserved surrounding spaces.
  * Healthy permanent dentition with good hygiene.

Exclusion Criteria:

* Patients will be excluded:

  * Who are taking drugs that affect bone metabolism and the inflammatory process (for example corticosteroids, bisphosphonates), who have used anti-inflammatory drugs or analgesics for less than 1 week since placing elastomeric separators.
  * Present general pathologies (craniofacial anomalies) and local ones (dental anomalies) that affect the result of the movement of the teeth,
  * Smokers, embarrassed, or breastfeeding women.
  * Allergic to paracetamol®
  * During the investigation, another different drug was used, which was made available by the investigators, and the patient was informed about this alteration.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
pain control after placement of elastomeric spacers - baseline | baseline
  Visual analogue scale
pain control after placement of elastomeric spacers - 24 hours | 24 hours
  Visual analog scale measuing 0 to 10 were "0" is no pain and "10" is the worst pain in life
pain control after placement of elastomeric spacers - 72 hours | 72 hours
  Visual analog scale measuing 0 to 10 were "0" is no pain and "10" is the worst pain in life

SECONDARY OUTCOMES:
Number of analgesics taken baseline | baseline
  The analgesic used will only be paracetamol. It will be used only if there is pain.
Number of analgesics taken 3 days | 3 days after procedure
  The analgesic used will only be paracetamol. It will be used only if there is pain.
Local temperature baseline | baseline
  evaluated using a digital thermometer
Local temperature 24 hours | 24 hours
  evaluated using a digital thermometer
The quality of life related to oral health baseline | baseline
  will be evaluated using the OHIP-14 questionnaire
The quality of life related to oral health -72 hours | 72 hours
  will be evaluated using the OHIP-14 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Carolina R.T. Horliana, São Paulo, São Paulo, Brazil